CLINICAL TRIAL: NCT01940978
Title: A Double-Blind Placebo-Controlled Study of Combination Therapy in Children With ADHD
Brief Title: A Study of Combination Therapy in Children With ADHD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Douglas Sears (Individual)
Responsible Party: Sponsor-Investigator, Douglas Sears, Douglas Sears, MD, Sears, Douglas, M.D.
Organization: Sears, Douglas, M.D. (Individual)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2013-09-09; First posted 2013-09-12 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: ADHD; Attention Deficit Hyperactivity Disorder; Attention Deficit Disorder With Hyperactivity; Mental Disorders Diagnosed in Childhood; Attention Deficit and Disruptive Behavior Disorders
Keywords: Methamphetamine; Methylphenidate; ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Neurodevelopmental Disorders; Attention Deficit and Disruptive Behavior Disorders | interventions — Methylphenidate; Cyproheptadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (Placebo Comparator): Methylphenidate ER QD placebo BID
  Interventions: Drug: Methylphenidate ER
- Methylphenidate ER, cyproheptadine 2.5mg (Active Comparator): Methylphenidate ER QD cyproheptadine hydrochloride 2.5mg BID
  Interventions: Drug: Methylphenidate ER; Drug: Cyproheptadine
- Methylphenidate ER, cyproheptadine 5mg (Active Comparator): Methylphenidate ER QD cyproheptadine hydrochloride 5.0mg BID
  Interventions: Drug: Methylphenidate ER; Drug: Cyproheptadine

INTERVENTIONS:
Drug: Methylphenidate ER — Watson generic, starting dose 18mg QD
  Other Names: Concerta
Drug: Cyproheptadine — cyproheptadine hydrochloride
  Other Names: Periactin
  Arms: Methylphenidate ER, cyproheptadine 2.5mg; Methylphenidate ER, cyproheptadine 5mg

SUMMARY:
Lack of appetite and weight loss are a common side effect of ADHD therapy with amphetamines such as methylphenidate. Lack of sufficient food intake has been shown to have negative effects on weight and height as well as learning and memory.

There is no current treatment to prevent this loss of appetite except discontinuation or reduction of the methylphenidate. Discontinuation or reduction of the drug can cause the return of ADHD symptoms.

The purpose of this study is to compare the effects, good and/or bad, of two doses of a drug, cyproheptadine, vs placebo to find out if cyproheptadine prevents the appetite suppression associated with methylphenidate.

ELIGIBILITY:
Inclusion Criteria:

* The subject and subject's parents speak English
* Child or adolescent patients, male or female outpatients, who are at least 6 years of age, but must not yet have reached their 13th birthday prior to Visit 1, when informed consent is obtained
* Patients must meet Diagnostic and Statistical Manual of Mental Disorders Fourth Edition (DSM-IV) diagnostic criteria for ADHD (any subtype) and score at least 1.5 standard deviations above the age norm for their diagnostic subtype using published norms for the Swanson, Nolan and Pelham Questionnaire: Attention-Deficit/Hyperactivity Disorder Subscale (SNAP-IV ADHD Subscale) score at both Visit 1 and 2
* Laboratory results, including serum chemistries, hematology, and urinalysis, must show no clinically significant abnormalities (clinically significant is defined as laboratory values requiring acute medical intervention, indicating a serious medical illness, or requiring further medical evaluation in the judgment of the investigator)
* Patients and parents have been judged by the investigator to be reliable to keep appointments for clinic visits and all tests, including venipuncture, and examinations required by the protocol.
* Patient has not been on stimulants for at least 2 weeks.

Exclusion Criteria:

* Patients who have a documented history of Bipolar I or II disorder, or any history of psychosis. Diabetic patients or patients on chronic steroids.
* Patients with a history of any seizure disorder (other than febrile seizures) or patients who have taken (or are currently taking) anticonvulsants for seizure control are not eligible to participate
* Patients at serious suicidal risk as defined by 1) suicidal ideation as endorsed on items 4 and 5 of the C-SSRS within the past year, 2) suicidal behaviors detected by the C-SSRS during the past two years; or 3) psychiatric interview and examination
* Patients with significant cardiovascular disease or other conditions that could be aggravated by an increased heart rate or increased blood pressure
* Patients who have any medical condition that would increase sympathetic nervous system activity markedly (for example, catecholamine-secreting neural tumor), or who are taking a medication on a daily basis (for example, albuterol, inhalation aerosols, pseudoephedrine), that has sympathomimetic activity. Such medications can be taken on an as-needed basis
* Presence of contraindications for methylphenidate or cyproheptadine hydrochloride
* Patients who have had prior serious adverse reaction to stimulants.
* Parental or (immediate) family history of substance abuse

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 99 (Actual)
Dates: Start 2014-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Appetite - Appetite and Dietary Assessment Tool (ADAT) developed by Burrowes et al (1996) | 0, 12 weeks

SECONDARY OUTCOMES:
Swanson, Nolan & Pelham Rating Scale - Revised (SNAP-IV): ADHD Combined Score | 0,1,5,9,12 weeks
  The items from the DSM-IV (1994) criteria for Attention-Deficit/Hyperactivity Disorder (ADHD) are included for the two subsets of symptoms: inattention (items #1-#9) and hyperactivity/ impulsivity (items #11-#19).
Weight | 0,1,5,9,12 Weeks
Appetite - VAS - Visual Analogue Scale | 0,1,5,9,12
Clinical Global Impressions - Improvement(CGI-I): ADHD Score | 1,5,9,12 weeks
Clinical Global Impressions - Severity(CGI-S): ADHD Score | 0,1,5,9,12
Clinical Global Impressions - Effectiveness(CGI-E): ADHD Score | 1,5,9,12
Appetite - Appetite and Dietary Assessment Tool (ADAT) developed by Burrowes et al (1996) | 1,5,9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Schuster, MD, Principal Investigator — SMRI
Locations (1):
- SMRI (Schuster Medical Research Institute), Van Nuys, California, United States